CLINICAL TRIAL: NCT02479867
Title: Comparative Open-label,Randomized, Fasting, Single Dose, Two-way Crossover Bioequivalence Study of Cefadroxil From Duricef 1 gm F.C.T (GSK) and Biodroxil 1 gm F.C.T (Novartis Pharma)
Brief Title: A Bioequivalence Study of Cefadroxil From Duricef 1 gm F.C.T (GSK) and Biodroxil 1 gm F.C.T (Novartis Pharma)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genuine Research Center, Egypt (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: GRC/1/13/515
Record Dates: First submitted 2015-06-15; First posted 2015-06-24 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
MeSH Terms: interventions — Cefadroxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A Test (Experimental): Test drug (Duricef) 1 tablet contains 1 gm Cefadroxil
  Interventions: Drug: Cefadroxil
- B Reference (Experimental): Reference drug (Biodroxil) 1 tablet contains 1 gm Cefadroxil
  Interventions: Drug: Cefadroxil

INTERVENTIONS:
Drug: Cefadroxil — 1 tablet from test vs 1 tablet from reference
  Other Names: Biodroxil

SUMMARY:
Comparative randomized, single dose, two-way crossover open-label study to determine the bioequivalence of Cefadroxil from Duricef 1 gm Film Coated tablets(Smthkline Beecham Egypt,LLC affiliated co. to GalaxoSmithKline ) and Biodroxil 1 gm Film Coated tablets (Kahira Pharm &Chem .Ind. Co . for Novartis Pharma ) after a single oral dose administration of each to healthy adults under fasting conditions.

DETAILED DESCRIPTION:
14 blood samples will be drawn in each period. The total volume of blood will not exceed 200 ml throughout the whole study. 0.00, 0.25, 0.50, 0.75, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00 and 12.00 hours., Primary Pharmacokinetic Parameters: Cmax, AUC0→t and AUC0→∞ Secondary Pharmacokinetic Parameters: Ke, tmax and t1/2e. ANOVAusing 5% significance level for transformed (with the 90% confidence intervals) and untransformed data of Cmax, AUC0→t and AUC0→∞ and for untransformed data of Ke, tmax and t1/2e.

The confidence intervals of logarithmically transformed Test/Reference ratios forCmax, AUC0→t and AUC0→∞ to be within 80.00-125.00%.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, age 18 to 55 years, inclusive.
2. Body weight within 15% of normal range according to the accepted normal values for body mass index (BMI)
3. Medical demographics without evidence of clinically significant deviation from normal medical condition.
4. Results of clinical laboratory test are within the normal range or with a deviation that is not considered clinically significant by principal investigator.
5. Subject does not have allergy to the drugs under investigation.

Exclusion Criteria:

1. Subjects with known allergy to the products tested.
2. Subjects whose values of BMI were outside the accepted normal ranges.
3. Female subjects who were pregnant, nursing or taking birth control pills.
4. Medical demographics with evidence of clinically significant deviation from normal medical condition.
5. Results of laboratory tests which are clinically significant.
6. Acute infection within one week preceding first study drug administration.
7. History of drug or alcohol abuse.
8. Subject does not agree not to take any prescription or non-prescription drugs within two weeks before first study drug administration and until the end of the study.
9. Subject is on a special diet (for example subject is vegetarian).
10. Subject does not agree not to consume any beverages or foods containing methyl-xanthenes e.g. caffeine (coffee, tea, cola, chocolate etc.) 48 hours prior to the study administration of either study period until donating the last sample in each respective period.
11. Subject does not agree not to consume any beverages or foods containing grapefruit 7 days prior to first study drug administration until the end of the study.
12. Subject has a history of severe diseases which have direct impact on the study.
13. Participation in a bioequivalence study or in a clinical study within the last 6 weeks before first study drug administration.
14. Subject intends to be hospitalized within 6 weeks after first study drug administration.
15. Subjects who, through completion of this study, would have donated more than 500 ml of blood in 7 days, or 750 ml of blood in 30 days, 1000 ml in 90 days, 1250 ml in 120 days, 1500 ml in 180 days, 2000 ml in 270 days, 2500 ml of blood in 1 year.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Maximal measured plasma concentration (Cmax) | 12 hours
  Serial blood samples for determination of study drug will be collected pre-dose and at 0.00 (pre-dose), 0.25, 0.50, 0.75, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00 and 12.00 hours.

SECONDARY OUTCOMES:
Time of the maximum plasma concentration (tmax)measurable concentration (t) | 12 hours
  The elimination or terminal half-life will be calculated as 0.693/ Ke

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elshafeey, Ph.D.Pharma, Study Director — ahmed.elshafeey@grc-me.com
Locations (1):
- Genuine Research Center GRC, Cairo, Egypt

REFERENCES:
- See also: International conference of Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use. ICH Harmonized Tripartite Guideline Q2B. Guidelines for Validation of Analytical Procedures: Methodology. November, 1996 — http://www.pharmaweb.net/pwmirror/pw9/ifpma/ICH1.html